CLINICAL TRIAL: NCT06874413
Title: Targeted Prehabilitation With Physical Exercise and Inspiratory Muscle Training for Elderly Frail Patients Prior to Ventral Hernia Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2290314
Record Dates: First submitted 2025-02-18; First posted 2025-03-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Frailty; Ventral Hernia
MeSH Terms: conditions — Frailty; Hernia, Ventral | interventions — Preoperative Exercise; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 - Standard of Care (Active Comparator): Patient receives standard of care instructions for preparing for ventral hernia repair surgery and recovery. Postoperative outcomes are measured.
  Interventions: Other: Standard of Care (SOC)
- Group 2 - Physical Exercise Arm (Experimental): Elderly patients with frailty participate in a 6-8 weeks of physical exercise program through the YMCA's SilverSneakers Program monitored by a wearable activity monitor. Patients will also complete respiratory training by using an incentive spirometer daily. Postoperative outcomes are measured
  Interventions: Behavioral: Prehabilitation
- Group 3 - Observational Cohort (No Intervention): Patient's physical activity is monitored prior to receiving ventral hernia repair surgery and postoperative outcomes are measured.

INTERVENTIONS:
Behavioral: Prehabilitation — Physical prehabilitation or exercise conducted through the YMCA's Silver Sneaker's program prior to receiving surgery that will be assessed through the use of wearable activity monitors.
  Arms: Group 2 - Physical Exercise Arm
Other: Standard of Care (SOC) — Patients will receive standard of care preoperative instructions.
  Arms: Group 1 - Standard of Care

SUMMARY:
The purpose of this study is to assess the physical fitness of patients undergoing hernia repair and correlate the postoperative outcomes and recovery as well as assess the impact of a targeted physical exercise program preoperatively in a cohort of frail, elderly patients.

The investigators hypothesize that physical exercise will improve activity levels in elderly patients with frailty prior to ventral hernia repair. The investigators further hypothesize that increased levels of activity preoperatively will correlate with improved postoperative outcomes.

DETAILED DESCRIPTION:
The goals of this study are to:

* assess the impact of a targeted physical exercise program on activity levels prior to ventral hernia repair in elderly, frail patients using wearable activity monitoring.
* correlate physical activity and the impact of physical exercise with postoperative outcomes, including quality of life, postoperative complications, length of hospital stay, discharge to home, and return to baseline activity.

The investigators intend to randomize one group of elderly, frail patients to perform an exercise program for 6-8 weeks prior to surgery and another group of elderly, frail patients to receive standard of care preoperative instructions.

The investigators will also collect data from a cohort of patients receiving a ventral hernia repair who have a wearable activity monitor that are willing to download an application on their phone and allow us to monitor their activity levels prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1 & 2:

  * Age 65 or greater
  * Presence of a ventral hernia with plans for elective hernia repair with mesh
  * Willing to consent to study and randomization, including activity data capture
  * Score of ≥6 and ≤11 on the Edmonton Frail Scale OR 5-item modified Frail Index Score > 0
  * For patients with cardiac disease, additional referral for cardiac risk assessment may be performed at the discretion of the treating surgeon or anesthesiologist. If deemed appropriate risk, patients may still enroll.
  * Uses a smartphone that is capable of downloading the Health Kit application
* Group 3:

  * Age 18 or older
  * Presence of a ventral hernia with plans for elective repair with mesh
  * Willing to consent to activity data capture
  * Uses a smartphone that is capable of downloading the Health Kit application

Exclusion Criteria:

* Group 1 &2:

  * Age <65
  * Unwilling or unable to consent to study or randomization
  * Joint or muscle pain with movement at a level of 5 out of 10 or higher per patient report
  * Score of ≤5 or ≥12 on Edmonton Frail Scale
  * mFI-5 positive for congestive heart failure (newly diagnosed or exacerbated within 30 days)
  * Functional dependence that prevents self-guided physical prehabilitation or other condition medically unsuitable for exercises (as determined by surgeon).
  * BMI >50
  * Parastomal hernia repair or repair without mesh
  * Plan for concurrent procedure

Group 3:

* <18 y/o
* Unwilling or unable to consent to study
* Joint or muscle pain with movement at a level of 5 out of 10 or higher per patient report
* BMI >50
* Parastomal hernia repair or repair without mesh
* Plan for concurrent procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Activity levels | 6-8 weeks preoperatively
  Amount of time spent active measured by data from wearable activity monitors

SECONDARY OUTCOMES:
Quality of Life Pre- and Postoperative Assessment | 14-30 days postoperatively
  Quality of life will be measured with the Hernia-Related Quality of Life Survey (HerQLes). This survey is a 12 question survey that measures how strongly the patient agrees or disagrees (strongly, moderately, and slightly agree or disagree) with the statement.
Quality of Life Pre- and Postoperative Outcomes | 14-30 days postoperatively
  Quality of life as measured by the Patient-Reported Outcome Measurement Information System (PROMIS-3).
Postoperative Outcomes - Surgical Complications | 14-30 days postoperatively
  Postoperative complications
Postoperative Outcomes - Length of Stay | 14-30 days postoperatively
  Number of days staying in the hospital prior to discharge
Postoperative Outcomes - Discharge Location | 14-30 days postoperatively
  Discharge location
Postoperative Outcomes - Return to Baseline | 14-30 days postoperatively
  Ability to return to baseline activity

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Warren, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No